CLINICAL TRIAL: NCT05753709
Title: Conventional Hand Sewn End-To-End Anastomosis Versus Side-To-Side Anastomosis for Stoma Reversal: A Randomised Clinical Trial
Brief Title: Conventional Hand Sewn End-To-End Anastomosis Versus Side-To-Side Anastomosis for Stoma Reversal: A Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sawai Mansingh Medical College (Other Government)
Responsible Party: Principal Investigator, Tanmay Agarwal, Junior Resident, Principal Investigator, Sawai Mansingh Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37/MC/EC/2021
Record Dates: First submitted 2023-02-13; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Stoma Ileostomy; Stoma Colostomy; Anastomosis; Ileus; Leak, Anastomotic; Bowel Obstruction
MeSH Terms: conditions — Ileus; Anastomotic Leak; Intestinal Obstruction

STUDY DESIGN:
Intervention Model Description: two groups in parallel: EE and SS, and another comparison with three arms: EE versus SS divided into two separate arms: SSSA and HSSA
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EE (Active Comparator): End-to-end anastomosis, done in a conventionally described hand-sewn technique using sutures
  Interventions: Procedure: Hand sewn end-to-end anastomosis
- SSSA (Active Comparator): Stapled side-to-side anastomosis of the stoma using a linear cutter stapling device
  Interventions: Procedure: Stapled side-to-side anastomosis
- HSSA (Active Comparator): Hand-sewn anastomosis of the stoma using suturing of bowel loops placed in a side to side orientation
  Interventions: Procedure: Hand sewn side-to-side anastomosis

INTERVENTIONS:
Procedure: Hand sewn end-to-end anastomosis — Hand sewn end-to-end anastomosis (EE) Holding sutures were taken through a seromuscular bite with PDS (Polydiaxonone) 3-0 or Silk 2-0 RB (Round Bodied needle), one each at the mesenteric and antimesenteric ends of the stoma. A posterior layer of Lembert sutures was taken first. The first bite was taken at the anti-mesenteric end and a knot was applied. A Connell stitch was applied at the corner and then the posterior layer was closed using an inverting interlocking continuous stitch till the mesenteric end. Another Connell stitch was applied here to secure the corner and the suture was continued on to the anterior layer which was then closed in a similar manner using a continuous interlocking stitch. The final bite crossed the initial knot and the final knot was applied. An anterior layer of Lembert sutures was taken to reinforce the anastomotic line.
  Arms: EE
Procedure: Hand sewn side-to-side anastomosis — Hand sewn side-to-side anastomosis (HSSA) Each end of the stoma was closed using either a single layer of inverting interlocking continuous sutures with PDS 3-0 or Silk 2-0 RB, or a Linear Stapling device. The two closed stumps were then brought adjacent to each other in an anti-peristaltic arrangement. A posterior layer of Lembert sutures was applied using Silk 2-0 RB. The bowel wall was incised using electrocautery close to the suture line. The incision was lengthened up to a width of at least 5-6 cm. The posterior and anterior layer was now closed using the same technique as in HS using PDS 3-0. An anterior layer of Lembert sutures was applied. The mesenteric defect was then closed using a superficial interrupted layer of Silk 2-0 RB.
  Arms: HSSA
Procedure: Stapled side-to-side anastomosis — Stapled side-to-side anastomosis or Functional End-to-end anastomosis (SSSA/FEEA) The two limbs of a Linear Cutter SR55 are placed into the proximal and distal bowel loops of the stoma, facing as far away from the mesenteric border as possible and then fired. If both lumens are of similar size, traction sutures are applied with Silk 2-0 RB at the anterior and posterior termination ends of the staple line. The two ends are pulled away from each other, and a Linear Cutter SR75 is applied just below the edge of the bowel and fired. However, in case of an ileo-colostomy, after the first linear cutter SR55 is fired, the two suture lines are approximated in such a way that they do not get apposed but rather lie adjacent to each other. The lumen is then clamped in SR75 which is then fired.
  Arms: SSSA

SUMMARY:
The goal of this clinical trial is to compare approaches to enterostomy reversal by hand-sewn end-to-end anastomosis versus side-to-side anastomosis (sub-divided into hand-sewn side-to-side anastomosis and stapled side-to-side anastomosis). The main question it aims to answer is:

• If either of the approaches are better than the other with respect to success rates, efficacy, post-operative complications and overall morbidity.

Participants admitted for stoma reversal will be divided into two groups:

1. EE: Conventional Hand-sewn end-to-end anastomosis, and
2. SS: Side-to-side anastomosis, which will be further divided into 2 sub-groups:

   1. HSSA: Hand-sewn side-to-side anastomosis
   2. SSSA: Stapled side-to-side anastomosis

Researchers will compare the EE group to SS group overall, and a second comparison will be made between EE, HSSA and SSSA groups, to see:

1. Rates of major post-operative complications
2. Rates of short-term complications (within 30 days of surgery)
3. Rates of re-operation
4. Post-operative length of stay in the hospital

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were all the patients admitted in general surgical wards of SMS Hospital, Jaipur, for stoma reversal, after taking written informed consent

Exclusion Criteria:

* Pre-operatively diagnosed malnutrition or cachexia
* Bleeding disorders
* Patients undergoing stoma reversal along with a concurrent abdominal surgery
* Rectal anastomosis
* Use of circular stapler for anastomosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with Post-operative Ileus (POI) | From the day of surgery for 30 days
  Number of participants with two or more episodes of nausea/vomiting, inability to tolerate oral diet over 24 hours, absence of flatus over 24 hours, or distension, and with radiologic confirmation, occurring postoperatively without spontaneous resolution
Number of participants with Anastomotic Leak | From the day of surgery for 30 days
  Number of participants with leakage of bowel contents from the anastomotic site, confirmed with imaging studies and clinical signs, such as fever >38.5˚C, leucocytosis, elevated serum C-reactive protein, drainage of intestinal content from the drain or computed tomography findings of abscess formation around the anastomosis.
Number of participants with complications of Clavien-Dindo grade higher than 2 | From the day of surgery for 30 days
  Number of participants with complications developing post-operatively of Clavien-Dindo grade higher than 2, suggestive of a severe complication.
Number of participants with Bowel Obstruction | From the day of surgery for 30 days
  Number of participants with Bowel dilatation and obstipation (inability to pass flatus as well as motion), requiring surgery for treatment, with transition point of the obstruction confirmed either radiologically or intraoperatively

SECONDARY OUTCOMES:
Operating Time | Intraoperatively
  Time during surgery from incision to skin closure
Number of participants with Wound Infection | From the day of surgery for 30 days
  Number of participants with Infection of the incision site ranging from simple local purulent collection to overt infection requiring re-operation
Number of participants with Anastomotic Bleeding | From the day of surgery for 30 days
  Number of participants with Evidence of bleeding around the anastomotic site, confirmed by a complaint of melena, or radiological or endoscopic findings.
Number of participants with Anastomotic Stricture | From the day of surgery for 30 days
  Number of participants with Imaging studies done in patients with complaints of nausea or bloating after oral intake, demonstrating intestinal distension starting from oral side of the anastomotic site, occurring due to narrowing at the site of anastomosis due to any cause. This did not include patients unable to pass flatus and motion (obstipation, criteria for bowel obstruction) or patients only unable to tolerate oral diet without other symptoms (criteria for POI).
Number of participants with Intra-abdominal Collection | From the day of surgery for 30 days
  Number of participants with fluid collection inside the abdominal cavity developing post-operatively, of any origin, which was not present before surgery. The fluid collection includes presence of ascitic fluid, blood or pus, in amount sufficient to be detected by an abdominal ultrasound or computed tomography imaging. The number of participants showing presence of fluid was measured, and not the volume of fluid.
Number of participants with Re-operation | From the day of surgery for 30 days
  Number of participants developing complications severe enough and not responding to medical management, that needed to be re-operated
Number of participants with Organ Dysfunction for each individual organ | From the day of surgery for 30 days
  Number of participants with Dysfunction in any organ, evidenced by symptoms and blood tests, developing post-operatively and not present before surgery. The outcome was measured as the number of participants developing dysfunction of each a particular organ system, labelled as Renal, Cardiac, Hepatic, Vascular and Respiratory.
Overall Morbidity | From the day of surgery for 30 days
  The overall morbidity is reflective of the number of patients who have at least 1 complication; that is, patients who have at least 1 complication were counted only once, and only their highest-grade complication was counted, graded on the Clavien-Dindo scale.

OTHER OUTCOMES:
Days to Bowel Movement | From the day of surgery for 30 days
  number of days for patient to first pass flatus or first stool after surgery
Days to Liquid diet | From the day of surgery for 30 days
  number of days for patient to be first started on and tolerate liquids given per-orally, without causing vomiting or abdominal distension
Days to Solid diet | From the day of surgery for 30 days
  number of days for patient to be first started on and tolerate progressively increasing semi-solid diet given per-orally, without causing vomiting or abdominal distension
Postoperative length of stay | From the day of surgery for 30 days
  Number of days for the patient to be discharged from the hospital without complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Sawai Mansingh Medical College and Hospital, Jaipur, Rajasthan, India

REFERENCES:
- [Background] Stedman's Medical Dictionary. 27th ed. Baltimore: Lippincott Williams & Wilkins; 2000.
- [Background] Turnbull RB, Weakley FL. St Louis: Mosby. Atlas of intestinal stomas. 1967;32-9.
- [Background] Dinc B, Ay N, Ciyiltepe H. Comparing methods of ileostomy closure constructed in colorectal surgery in Turkey. Prz Gastroenterol. 2014;9(5):291-6. doi: 10.5114/pg.2014.46165. Epub 2014 Oct 19. PMID 25396004
- [Background] Prassas D, Ntolia A, Spiekermann JD, Rolfs TM, Schumacher FJ. Reversal of Diverting Loop Ileostomy Using Hand-Sewn Side-to-Side versus End-to-End Anastomosis after Low Anterior Resection for Rectal Cancer: A Single Center Experience. Am Surg. 2018 Nov 1;84(11):1741-1744. PMID 30747626
- [Background] Steichen FM. The use of staplers in anatomical side-to-side and functional end-to-end enteroanastomoses. Surgery. 1968 Nov;64(5):948-53. No abstract available. PMID 5687844
- [Background] Liu Z, Wang G, Yang M, Chen Y, Miao D, Muhammad S, Wang X. Ileocolonic anastomosis after right hemicolectomy for colon cancer: functional end-to-end or end-to-side? World J Surg Oncol. 2014 Oct 7;12:306. doi: 10.1186/1477-7819-12-306. PMID 25287418
- [Background] Sameshima S, Koketsu S, Yoneyama S, Miyato H, Kaji T, Sawada T. Outcome of functional end-to-end anastomosis following right hemicolectomy. Int Surg. 2009 Jul-Sep;94(3):249-53. PMID 20187520
- [Background] Goto T, Kawasaki K, Fujino Y, Kanemitsu K, Kamigaki T, Kuroda D, Suzuki Y, Kuroda Y. Evaluation of the mechanical strength and patency of functional end-to-end anastomoses. Surg Endosc. 2007 Sep;21(9):1508-11. doi: 10.1007/s00464-006-9131-6. Epub 2007 Feb 7. PMID 17285383
- [Background] Choy PY, Bissett IP, Docherty JG, Parry BR, Merrie A, Fitzgerald A. Stapled versus handsewn methods for ileocolic anastomoses. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD004320. doi: 10.1002/14651858.CD004320.pub3. PMID 21901690
- [Background] Loffler T, Rossion I, Goossen K, Saure D, Weitz J, Ulrich A, Buchler MW, Diener MK. Hand suture versus stapler for closure of loop ileostomy--a systematic review and meta-analysis of randomized controlled trials. Langenbecks Arch Surg. 2015 Feb;400(2):193-205. doi: 10.1007/s00423-014-1265-8. Epub 2014 Dec 25. PMID 25539702
- [Background] Loffler T, Rossion I, Bruckner T, Diener MK, Koch M, von Frankenberg M, Pochhammer J, Thomusch O, Kijak T, Simon T, Mihaljevic AL, Kruger M, Stein E, Prechtl G, Hodina R, Michal W, Strunk R, Henkel K, Bunse J, Jaschke G, Politt D, Heistermann HP, Fusser M, Lange C, Stamm A, Vosschulte A, Holzer R, Partecke LI, Burdzik E, Hug HM, Luntz SP, Kieser M, Buchler MW, Weitz J; HASTA Trial Group. HAnd Suture Versus STApling for Closure of Loop Ileostomy (HASTA Trial): results of a multicenter randomized trial (DRKS00000040). Ann Surg. 2012 Nov;256(5):828-35; discussion 835-6. doi: 10.1097/SLA.0b013e318272df97. PMID 23095628
- [Background] Chassin JL, Rifkind KM, Turner JW. Errors and pitfalls in stapling gastrointestinal tract anastomoses. Surg Clin North Am. 1984 Jun;64(3):441-59. doi: 10.1016/s0039-6109(16)43330-x. PMID 6379923
- [Background] Perez RO, Habr-Gama A, Seid VE, Proscurshim I, Sousa AH Jr, Kiss DR, Linhares M, Sapucahy M, Gama-Rodrigues J. Loop ileostomy morbidity: timing of closure matters. Dis Colon Rectum. 2006 Oct;49(10):1539-45. doi: 10.1007/s10350-006-0645-8. PMID 16897328
- [Background] Flikier-Zelkowicz B, Codina-Cazador A, Farres-Coll R, Olivet-Pujol F, Martin-Grillo A, Pujadas-de Palol M. [Morbidity and mortality associated with diverting ileostomy closures in rectal cancer surgery]. Cir Esp. 2008 Jul;84(1):16-9. doi: 10.1016/s0009-739x(08)70598-0. Spanish. PMID 18590670
- [Background] Hiranyakas A, Rather A, da Silva G, Weiss EG, Wexner SD. Loop ileostomy closure after laparoscopic versus open surgery: is there a difference? Surg Endosc. 2013 Jan;27(1):90-4. doi: 10.1007/s00464-012-2422-1. Epub 2012 Jun 30. PMID 22752281
- [Background] Klink CD, Wunschmann M, Binnebosel M, Alizai HP, Lambertz A, Boehm G, Neumann UP, Krones CJ. Influence of skin closure technique on surgical site infection after loop ileostomy reversal: retrospective cohort study. Int J Surg. 2013;11(10):1123-5. doi: 10.1016/j.ijsu.2013.09.003. Epub 2013 Sep 12. PMID 24035923
- [Background] Livingston EH, Passaro EP Jr. Postoperative ileus. Dig Dis Sci. 1990 Jan;35(1):121-32. doi: 10.1007/BF01537233. PMID 2403907
- [Background] Leung TT, MacLean AR, Buie WD, Dixon E. Comparison of stapled versus handsewn loop ileostomy closure: a meta-analysis. J Gastrointest Surg. 2008 May;12(5):939-44. doi: 10.1007/s11605-007-0435-1. Epub 2007 Dec 11. PMID 18071833
- [Background] Kaidar-Person O, Person B, Wexner SD. Complications of construction and closure of temporary loop ileostomy. J Am Coll Surg. 2005 Nov;201(5):759-73. doi: 10.1016/j.jamcollsurg.2005.06.002. Epub 2005 Sep 6. No abstract available. PMID 16256921
- [Background] Fauno L, Rasmussen C, Sloth KK, Sloth AM, Tottrup A. Low complication rate after stoma closure. Consultants attended 90% of the operations. Colorectal Dis. 2012 Aug;14(8):e499-505. doi: 10.1111/j.1463-1318.2012.02991.x. PMID 22340709
- [Background] Nagell CF, Pedersen CR, Gyrtrup HJ. [Complications after stoma closure. A retrospective study of 11 years' experience]. Ugeskr Laeger. 2005 Apr 18;167(16):1742-5. No abstract available. Danish. PMID 15898604
- [Background] Baastrup NN, Hartwig MFS, Krarup PM, Jorgensen LN, Jensen KK. Anastomotic Leakage After Stoma Reversal Combined with Incisional Hernia Repair. World J Surg. 2019 Apr;43(4):988-997. doi: 10.1007/s00268-018-4866-5. PMID 30483884
- [Background] Zarnescu EC, Zarnescu NO, Costea R. Updates of Risk Factors for Anastomotic Leakage after Colorectal Surgery. Diagnostics (Basel). 2021 Dec 17;11(12):2382. doi: 10.3390/diagnostics11122382. PMID 34943616